CLINICAL TRIAL: NCT00740766
Title: Perinatal Outcomes in Nutritionally Monitored Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamaica Hospital Medical Center (Other)
Responsible Party: Yvonne S. Thornton, M. D., M. P. H., New York Medical College
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#02-017; MMH IRB#R98-05-022; SLRHC IRB#01-138
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Obesity
Keywords: Perinatal Outcomes; Obesity; Pregnant women
MeSH Terms: conditions — Obesity | interventions — Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitored (Experimental)
  Interventions: Behavioral: Food diary and behavioral model
- Unmonitored (No Intervention)

INTERVENTIONS:
Behavioral: Food diary and behavioral model — The monitored group is to be placed on a prenatal nutritional program consisting of 18 to 24 kcal. per kg. (according to the patient's actual weight) with monitoring each visit.
  The patients will be weighed each prenatal visit with the monitored patients weighed and blinded to their actual weight (being weighed with her back to the scale). The monitored patients will be requested not to weigh at home and all patients will be asked to wear similar clothing at each visit.
  All intervention (monitored) group women will be asked to record in a diary all of the foods eaten during each day. These records will be reviewed at each prenatal visit. Six weeks after delivery, the patient will be weighed and will then exit the study. The food diary notebooks will be collected from each patient at the end of the study.
  Other Names: Adherence to prenatal nutritional program
  Arms: Monitored

SUMMARY:
The aim of this prospective randomized study is the prevention of excessive weight gain in obese pregnant women. The study will compare perinatal outcomes of obese pregnant women treated in the traditional way to outcomes of nutritionally monitored obese pregnant women and evaluate a preliminary behavioral model applicable to the general practice of obstetrics.

DETAILED DESCRIPTION:
Study Population and Selection:

This study will recruit 200 obese pregnant women at 12 to 28 weeks of gestation with a body mass index (BMI) of greater than 29.9 kg/m2. Women will be eligible if they are pregnant with a single fetus, and are free of diabetes, hypertension, or chronic kidney disease at recruitment.

Methodology:

The patients will be randomized to either traditional or monitored groups. All participants will be counseled at least once regarding conventional prenatal nutrition guidelines. A more detailed dietary intake protocol would be done with the intervention (monitored) group, which would include being placed on a balanced nutritional intake regimen of 18-24 kcal/kg/day (no less than 2000 calories). Each patient will be asked to record in a diary all of the foods she eats during the day, which will be reviewed by the investigator or assignee at each prenatal visit. The patients will be weighed at each prenatal visit with the monitored patients weighed and blinded to their actual weight.

Data analysis:

The two groups will be compared with respect to pregnancy weight gain, proportion of excessive weight gain (greater than 15 pounds), maternal morbidity, intrapartum complications and newborn birthweight. The primary analysis will consist of a two sample t-test comparing the monitored versus non-monitored groups with regard to weight gain at delivery. A secondary analysis using a repeated measures ANOVA will look at weight gain in the two groups from baseline to 6 weeks post partum in order to look at trends over time. Tests of mean contrasts will compare differences between the two groups at each time during and post pregnancy relative to baseline. Additional analyses will be done to look at other outcomes. In the case of continuous variable outcomes (e.g., gestational weight), a student's t-test will be used. while for categorical outcomes (e.g., macrosomia), the chi square test will be used for the comparison. Alpha will be 0.05 for each comparison.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 29.9 kg/m2
* Single fetus

Exclusion Criteria:

* Diabetes
* Hypertension or chronic kidney disease

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 1998-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Mean weight gain Proportion with excessive weight gain (greater than 15 pounds) Mean postpartum weight increment Newborn birthweight and length, controlled for gestational age Proportion of macrosomia Incidence of co-morbidities | From entry until 6-weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne S Thornton, MD, MPH, Principal Investigator
Locations (3):
- United States (3):
  - Morristown Memorial Hospital, Morristown, New Jersey
  - St. Luke's-Roosevelt Hospital, New York, New York
  - Jamaica Hospital Medical Center, New York, New York

REFERENCES:
- [Result] Thornton YS, Smarkola C, Kopacz SM, Ishoof SB. Perinatal outcomes in nutritionally monitored obese pregnant women: a randomized clinical trial. J Natl Med Assoc. 2009 Jun;101(6):569-77. doi: 10.1016/s0027-9684(15)30942-1. PMID 19585925